CLINICAL TRIAL: NCT03798834
Title: Fascia Iliaca Block as an Anesthetic Technique for Thromboembolectomy of Chronic Lower Limb Ischemia
Brief Title: Fascia Iliaca Block for Anesthesia in Lower Limb Thromboembolectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R/17.07.111
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Chronic Lower Limb Ischemia
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia iliaca block (FIB) (Experimental): ultrasound-guided Fascia iliaca block
  Interventions: Drug: Fascia iliaca block (FIB)
- Spinal anesthesia (Placebo Comparator): Spinal anaesthesia using 2 ml hyperbaric bupivacaine 0.5%
  Interventions: Other: Spinal anesthesia

INTERVENTIONS:
Drug: Fascia iliaca block (FIB) — ultrasound-guided Fascia iliaca block
  Arms: Fascia iliaca block (FIB)
Other: Spinal anesthesia — Spinal anaesthesia using 2 ml hyperbaric bupivacaine 0.5%
  Arms: Spinal anesthesia

SUMMARY:
The fascia iliaca block (FIB) is an anterior approach to block the lumbar plexus. It disturbed mainly to the anterior region of the thigh by blocking the femoral nerve (LFC) and the lateral femoral cutaneous nerve. Moreover, FIB may possibly be extended to the obturator, ilioinguinal, genitofemoral, lateral cutaneous nerve of the thigh and over the psoas muscle but, rarely reaches the lumbar plexus.

The fascia iliaca compartment could be detected by bony landmarks palpation and the loss of resistance technique. Feeling two tactile ''pops'' due to loss of resistance occurred during the needle passage through the fascia lata and the fascia iliaca. Ultrasound (US) guidance of FIB will increase the success rate and the efficacy of sensory blockade by decreasing the needed local anesthetic amount.

DETAILED DESCRIPTION:
This study was conducted to demonstrate the success incidence (to evaluate the efficacy) of preoperative 0.25% bupivacaine FIB as a sole anesthetic technique in thromboembolectomy of unilateral chronic lower limb ischemia compared to neuraxial anesthesiaas a primary goal. Intraoperative hemodynamics variation, postoperative pain score, total analgesic rescue requests and the total amount of systemic rescue analgesia used in the first postoperative day in addition to any detected postoperative complications were secondary goals. The hypothesis is that; FIB will provide adequate anesthesia as neuraxial anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II.

Exclusion Criteria:

* Patients with previous same lower limb surgery
* Neuromuscular disease
* Severe cardiovascular disease
* Any contraindications to regional anesthesia
* patient refusal
* coagulation abnormality
* Known allergy to local anesthetics
* Infection at the injection site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-11-17 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
The proportion of the patients who did not require conversion to general anesthesia | for 30 minutes

SECONDARY OUTCOMES:
Postoperative pain | For 24 hours after the intervention
  The post-operative pain will recorded using 10-point Visual Analog Scale (VAS)
Heart rate | For 6 hours after the intervention
  changes in Heart rate
mean arterial pressure (MAP | For 6 hours after the intervention
  changes in mean arterial pressure (MAP
hypotension | For 24 hours from the block
  Incidents of hypotension
Any observed adverse effects | over the 24 hours postoperative
  ny adverse effects will be observed over the 24 hours postoperative for local skin hematoma ,sensory deficits or local bleeding
bradycardia | For 24 hours from the block
  Incidents if bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Reem A Elsharkawy, MD, Study Chair — Lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided